CLINICAL TRIAL: NCT05124132
Title: Resilience and Brain Health of Older Adults (MEDEX-2)
Acronym: MEDEX-2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of California, San Diego (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 201810006; 1R01AG072694-01A1 (NIH)
Record Dates: First submitted 2021-11-15; First posted 2021-11-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Age-related Cognitive Decline
Keywords: Exercise; Mindfulness; Education; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness-Based Stress Reduction; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness-Based Stress Reduction (Experimental): Mindfulness-Based Stress Reduction (MBSR) as delivered in the parent study (Protocol ID #201410093) consisted of a brief introductory meeting, eight weekly 2.5-hour classes, and a retreat, followed by monthly booster sessions for approximately 15 months. Content included instruction in mindfulness meditation practices, gentle mindful movement, and exercises to enhance mindfulness in everyday life. For the current study, participants will continue monthly approximately 2.5 hour booster sessions covering similar content for the duration of the study. Participants will be encouraged to maintain daily formal meditative activities at home.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Exercise (Experimental): The exercise protocol in the parent study (Protocol ID #201410093) was optimal for improving aerobic fitness and insulin sensitivity in older adults, as well as improving strength and balance and reducing indices of frailty. It consisted of classes twice weekly for 6 months, building up to 1.5 hr, under the direct supervision of trained exercise instructors, followed by once weekly classes for 12 months. For the current study, participants will continue monthly approximately 1.5 hour classes focused on functional training for the duration of the study. Participants will be encouraged to continue between-session engagement in aerobic and resistance training activities at home.
  Interventions: Behavioral: Exercise
- Mindfulness-Based Stress Reduction + Exercise (Experimental): This condition will receive both MBSR and exercise as described. Participants in this condition will attend monthly sessions with encouragement to complete at-home mindfulness practice as well as at-home exercise for the duration of the study.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction + Exercise
- Health Education (Active Comparator): The health education control condition is based on a chronic disease self-management program developed at Stanford University and was used as an attentional control in the parent study (Protocol ID #201410093). This control intervention was designed to be time-equivalent to MBSR, with 8 weeks of 2.5 hour weekly group classes followed by monthly booster sessions for approximately 15 months. For the current study, participants will continue monthly approximately 1.5 hour sessions covering similar content for the duration of the study.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Mindfulness-Based Stress Reduction
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Exercise — Exercise
  Arms: Exercise
Behavioral: Mindfulness-Based Stress Reduction + Exercise — Mindfulness-Based Stress Reduction + Exercise
  Arms: Mindfulness-Based Stress Reduction + Exercise
Behavioral: Health Education — Health Education
  Arms: Health Education

SUMMARY:
This project capitalizes on a natural experiment imposed by the COVID-19 pandemic in conjunction with an extensive set of cognitive, emotional, biological, and neuroimaging variables already collected at multiple time points in older adults participating in a clinical trial of exercise and mindfulness. This project will elucidate the effects of stress on cognitive function and emotional health in later life, including biological measures of Alzheimer Disease risk, stress, and aging, with the ultimate goal of discovering how to mitigate these effects, among older adults who have made and maintained a lifestyle change.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the parent study, Protocol ID #201410093

Exclusion Criteria:

* Inability to safely continue classes or complete assessments, as per PI discretion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Effects of the interventions on changes in cognitive performance | Approximately three years
  Test effects of mindfulness and exercise on changes in change in memory and cognitive control composites.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact PI. Estimated date of availability December 2026.

REFERENCES:
- See also: Visit the Healthy Mind Lab for more information about the MEDEX study and our other areas of research. STL: http://healthymind.wustl.edu/medex UCSD: http://www.medexstudy.com/ — http://healthymind.wustl.edu/medex